CLINICAL TRIAL: NCT00696930
Title: A Phase II Open-label Multi-center Study to Evaluate the Efficacy and Safety of 90Y-SMT487 in Subjects With Symptomatic Malignant Carcinoid Tumors
Brief Title: Study to Evaluate the Efficacy and Safety of 90Y-SMT487 in Subjects With Symptomatic Malignant Carcinoid Tumors
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Molecular Insight Pharmaceuticals, Inc. (Industry)
Responsible Party: Molecular Insight Pharmaceuticals, Inc.
Purpose: Treatment
Other Study IDs: CSMT 487A 2202
Record Dates: First submitted 2008-06-11; First posted 2008-06-13 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2015-11

CONDITIONS: Malignant Carcinoid Tumor
Keywords: Malignant Carcinoid Tumors

INTERVENTIONS:
Drug: 90Y-SMT487

SUMMARY:
Subjects will be screened to determine OctreoScan® uptake. And upon meeting the eligibility criteria, 90 subjects will complete a symptom assessment scale at baseline and throughout the study at specific time points. Actual treatment will consist of three six-week cycles of a fixed total dose of 13.3 GBq (360 mCi) of 90Y-SMT487. The total dose will be divided into three equal doses and administered as a single activity of 4.4 GBq (120 mCi) of 90Y-SMT487 once every six weeks for three cycles. An amino acid infusion will be administered along with each dose. Long-term follow up will occur at 6 and 12 months after Day 1/ Cycle 1. Survival will be assessed every six months.

ELIGIBILITY:
Inclusion Criteria:

1. Life expectancy > 6 months.
2. Subjects must have distant metastases.
3. Subjects must be able to discontinue Sandostatin LAR treatment for at least 1 month prior to Day 1/Cycle 1; last dose of Sandostatin LAR must be 60 days or more prior to the first OctreoTher™ dose. For subcutaneous Sandostatin discontinuation should be 12 hours. Subjects taking other long acting somatostatin analogues must discontinue the analogue at least 2 times the dosing interval.
4. Upon baseline disease assessment, all subjects must have at least 1 measurable site of disease that either has never been irradiated or if the measurable lesion has been previously irradiated; this same lesion has since demonstrated progression base don the SWOG response criteria.
5. Subjects must state or agree with the statement that "I have symptoms from my cancer that bother me." Subjects must have failed to gain complete symptom control despite an optimal attempt at somatostatin therapy in the judgement of their physician.

Exclusion Criteria:

1. Chemotherapy, biologic therapy or other investigational therapy within 4 weeks of Day 1.
2. Surgery, hormonal therapy (not including somatostatin analogues) or radiation, within 2 weeks of Day 1.
3. Subjects with know brain metastases unless these metastases have been treated and stabilized for at least six months prior to study start.
4. Subjects who received high dose OctreoScan therapy or other radiolabelled somatostatin therapy or other systemic radiolabelled therapy (e.g. MIBG) for treatment of metastatic carcinoid.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-06; Primary Completion 2008-06 (Actual)